CLINICAL TRIAL: NCT00979186
Title: A Trial to Evaluate Natural Orifice Transgastric Endoscopic Cholecystectomy With Laparoscopic Assistance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Terminated - No enrollment, business decision.
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-08-0005
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2010-12

CONDITIONS: Cholecystectomy
Keywords: transgastric cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NOTES GEN 1 Toolbox — Articulating Hook Knife, Articulating Snare, Articulating Needle Knife Articulating Graspers, Articulating Biopsy Forceps, Steerable Flex Trocar with Rotary Access Needle, Flexible Bipolar Hemostasis Forceps, Flexible Maryland Dissector, and Tissue Apposition System.
  Other Names: Articulating Hook Knife, Articulating Snare, Articulating Needle Knife; Articulating Graspers, Articulating Biopsy Forceps, Steerable Flex Trocar with Rotary Access Needle,; Flexible Bipolar Hemostasis Forceps, Flexible Maryland Dissector, and Tissue Apposition System.

SUMMARY:
The study will document being able to successfully perform transgastric cholecystectomy (laparoscopic visualization) using a small collection of study surgical tools.

ELIGIBILITY:
Inclusion Criteria:

Men and women will be enrolled in this study who:

* Are willing to give consent and comply with evaluation and treatment schedule, able to understand and complete study questionnaires;
* At least 18 years of age;
* Have a clinical diagnosis of gallbladder disease indicated for cholecystectomy;
* ASA Classification I or II (Appendix II); and
* Have a negative serum pregnancy test (for women of childbearing potential);
* Have the study procedure attempted.

Exclusion Criteria:

* BMI > 35;
* Use of immunosuppressive medications (within 6 months of surgery; single burst dosages and inhalable steroids are acceptable);
* Suspicion of gallbladder cancer, tumor, polyps, or mass;
* Acute cholecystitis or acute pancreatitis;
* Presence of common bile duct stones;
* History of open abdominal surgery;
* Evidence of abdominal abscess or mass;
* Diffuse peritonitis;
* Use of anticoagulants or anti-platelet agents (use of daily cardio protective doses of aspirin, up to 81 mg/day, is acceptable and shall not constitute an exclusion criterion) or the presence of coagulopathy;
* Clinical diagnosis of sepsis;
* History of peritoneal trauma;
* Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or that could impact the scientific integrity of the trial;
* Planned concurrent surgical procedure;
* Prior or planned major surgical procedure within 30 days before or after study procedure;
* Previous diagnosis of intra-abdominal adhesions;
* Participation in any other investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints;
* Previously enrolled in the current series of 4 trials investigating the EES NOTES GEN1 Toolbox; or
* Any condition which precludes compliance with the study (Investigator discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proportion of procedures completed | 1 Day
  Day of surgery only - study complete at end of prodecure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, UCSD, San Diego, California, United States